CLINICAL TRIAL: NCT01590979
Title: Randomized Double Blind Control Trial on Effects of Ranolazine on New Onset Atrial Fibrillation Rates in Post-Operative Cardiac Surgery Patients
Brief Title: Randomized Double Blind Control Trial on Effects of Ranolazine on New Onset Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to slow rate of accrual resulting in a sample size.
Sponsor: Northwell Health (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Soad Bekheit, Director of Electrophysiology Lab, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bekheit-Ranolazine
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation New Onset; Hemorrhage; Prolonged QTc Interval; Ventricular Tachycardia; Medical Care; Complications, Late Effect of Complications
Keywords: Atrial Fibrillation New Onset; Ranolazine; CABG; valve repair/replacement; Cardiac Surgery
MeSH Terms: conditions — Hemorrhage; Tachycardia, Ventricular | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Active Comparator): The antianginal properties of the drug are due to inhibition of the late inward sodium current, demonstrated in animal experiments and human studies that it can prevent atrial and ventricular arrhythmias.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Company generated placebo, will be similar in size and color to Ranolazine; and administered two times a day (12 hour intervals)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 1000mg, two times a day, 12 hour intervals
  Other Names: RANEXA®
  Arms: Ranolazine
Drug: Placebo — two times a day, 12 hour intervals
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the prophylactic effects of Ranolazine on new onset atrial fibrillation in post-operative coronary artery bypass graft and valve surgery patient population at Staten Island University hospital.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common complication of cardiac surgery. It has been shown that the onset of AF increases in post-operative cardiac surgery population. The rate of AF after coronary artery bypass graft (CABG) procedure range from 10-65% and from 37-50% after valve surgery. Rates of new onset AF are lower for CABG compared to valve procedures. The pathophysiology of post-operative AF is not well elucidated. It has been postulated that pre-operative factors such as age, past medical history, operative and post-operative remodeling of the coronary system and hemodynamic pressure changes may contribute to post-operative AF.

Ranolazine is currently approved as an antianginal drug. The antianginal properties of the drug are due to inhibition of the late inward sodium current. Through the same mechanism it has been demonstrated in animal experiments and human studies that it can prevent atrial and ventricular arrhythmias.

Therefore it is important to prevent or minimize the incidence of new onset post-operative AF in post-surgical population.

ELIGIBILITY:
Inclusion criteria:

* Male and female candidates (18 years of age and older) undergoing coronary bypass grafting surgery or valve repair or replacement - Aortic or Tricuspid or Pulmonary valves
* Patients who are not previously on Ranolazine
* Do not have a history of arrhythmia and are not on any antiarrhythmic therapy
* Patients with QTc on a 12 lead EKG of less than or equal to 460 ms
* Patients with estimated Glomerular Filtration Rate (GFR) greater than 30 mL/min/1.73 m2 on the initial lab work
* Available at least 48 hours before surgery

Exclusion criteria:

* Patients who are not undergoing above surgeries
* Patients undergoing surgery for mitral valve replacement/repair
* Patient with cirrhosis
* Pregnant patients
* Patients with chronic atrial fibrillation
* Patients who had prior adverse drug reactions or allergies to Ranolazine
* Patients who are already taking Ranolazine prior to the study
* Patient who are reported HIV Positive (as there are antiretroviral drug interactions)
* Patients who are on drugs listed in Appendix A prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soad Bekheit, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hosptial, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The conversion of paroxysmal or initial onset atrial fibrillation with oral Ranolazine: Implications for a new "pill-in-pocket" approach in structural heart disease. — http://preview.ncbi.nlm.nih.gov/pubmed?term=Murdock%20DK%2C%20Kersten%20M%2C%20Kaliebe%20J%2C%20Larrain%20G
- See also: Comparison of effectiveness and safety of Ranolazine versus amiodarone for preventing atrial fibrillation after coronary artery bypass grafting. — http://preview.ncbi.nlm.nih.gov/pubmed?term=21726841
- See also: Electrophysiologic basis for the antiarrhythmic actions of Ranolazine. Heart Rhythm. — http://preview.ncbi.nlm.nih.gov/pubmed?term=21421082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (11.7) | 62.9 (11.1) | 64.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Incidence of New Onset Atrial Fibrillation Rate in Post-Operative Cardiac Surgery Patients
Time Frame: 3 weeks after surgery
Population: Fifty-four patients were randomized with a mean follow-up of 25 months and none were lost to follow-up. The study was terminated due to slow rate of accrual resulting in a sample size of 27 ranolazine and 27 placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 27 | 27
Participants | 5 | 8

ADVERSE EVENTS:
Time Frame: Post op (days 1-6); hospital discharge; Post -op follow up (2-3 weeks); Follow up call (day 28).
Description: Patients were given a medication log post discharge to note when medication was taken and to note any other comments related to how they were feeling.
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 4/27 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=27) | Placebo (N=27)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to insufficient accrual rate the study was stopped before the recruitment total was met. Thus, a major limitation is small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes